CLINICAL TRIAL: NCT06463392
Title: Development of Deep-Learning-Based Multimodal Post Radiotherapy Skull-Base Osteonecrosis and Recurrence of Nasopharyngeal Carcinoma Differential Diagnostic Model
Brief Title: Deep Learning-based sbORN Diagnostic Model
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-395-03
Record Dates: First submitted 2024-05-22; First posted 2024-06-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma; Herpesvirus 4, Human
Keywords: Nasopharyngeal Carcinoma; Skull-base Osteonecrosis; Radiotherapy; Epstein-Barr Virus
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Histologically confirmed sbORN that meets the eligibility criteria.
  Interventions: Other: No Intervention: Observational Cohort
- Control: Histologically confirmed NPC recurrence that meets the eligibility criteria.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention is scheduled for this observational study.

SUMMARY:
Skull-base osteonecrosis (sbORN) is a severe long-term complication of nasopharyngeal carcinoma (NPC) post radiotherapy, which significantly diminish the quality of life, increase the risk of internal carotid artery rupture, and is frequently misdiagnosed as NPC recurrence. Novel diagnostic tools are therefore clinically significant. In this study, the investigators seek to ask if a deep-learning-based model shows a significantly higher sensitivity than radiologists. With a cross-sectional design, the investigators aim to recruit 312 participants in Sun Yat-sen Memorial Hospital, Guangzhou, China that meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or older than 18 years old.
* A history of histologically confirmed nonkeratinizing undifferentiated nasopharyngeal carcinoma.
* A history of radical radiotherapy at nasopharynx.
* Complete remission six months post radical radiotherapy according to RECIST 1.1.
* No evidence of distant metastasis upon recruitment.
* Diagnosis of sbORN given by senior radiologist with 2-4 Likert scores.
* Consent to biopsy awake or under general anesthesia.
* Consent to perform blood tests, EBV DNA, EBV IgAs, and MRI inspection of nasopharynx and neck.
* With a written consent.

Exclusion Criteria:

* MRI artifacts or other factors that interfere radiological diagnosis and region of interest contouring.
* Suspected lesion is not confined to nasopharynx and skull-base.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All populations that meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under curve of the differential diagnosis of sbORN and NPC recurrence delivered by the deep-learning-based multimodal model. | Baseline
Area under curve of the differential diagnosis of sbORN and NPC recurrence delivered by the radiologists. | Baseline

SECONDARY OUTCOMES:
Sensitivity of the differential diagnosis of sbORN and NPC recurrence delivered by the deep-learning-based multimodal model. | Baseline
Specificity of the differential diagnosis of sbORN and NPC recurrence delivered by the deep-learning-based multimodal model. | Baseline
F1 score of the differential diagnosis of sbORN and NPC recurrence delivered by the deep-learning-based multimodal model. | Baseline
Positive predictive value of the differential diagnosis of sbORN and NPC recurrence delivered by the deep-learning-based multimodal model. | Baseline
Negative predictive value of the differential diagnosis of sbORN and NPC recurrence delivered by the deep-learning-based multimodal model. | Baseline
Sensitivity of the differential diagnosis of sbORN and NPC recurrence delivered by the radiologists. | Baseline
Specificity of the differential diagnosis of sbORN and NPC recurrence delivered by the radiologists. | Baseline
F1 score of the differential diagnosis of sbORN and NPC recurrence delivered by the radiologists. | Baseline
Positive predictive value of the differential diagnosis of sbORN and NPC recurrence delivered by the radiologists. | Baseline
Negative predictive value of the differential diagnosis of sbORN and NPC recurrence delivered by the radiologists. | Baseline
Dice similarity coefficient of the MRI contouring between the deep-learning-based multimodal model and the radiologists. | Baseline
Average surface distance of the MRI contouring between the deep-learning-based multimodal model and the radiologists. | Baseline

OTHER OUTCOMES:
The number of white blood cells in the peripheral blood. | Baseline
The number of neutrophils in the peripheral blood. | Baseline
The number of basophils in the peripheral blood. | Baseline
The number of eosinophils in the peripheral blood. | Baseline
The number of red blood cells in the peripheral blood. | Baseline
The concentration of albumin in the peripheral blood. | Baseline
The concentration of total protein in the peripheral blood. | Baseline
The history of diabetes mellitus. | Baseline
The history of hypertension. | Baseline
The copy number of Epstein-Barr Virus (EBV) DNA. | Baseline
The titer of EBV VCA IgA. | Baseline
The titer of EBV EBNA1 IgA. | Baseline
The titer of EBV EA IgA. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China